CLINICAL TRIAL: NCT01486108
Title: Burst, Tonic and Sham Spinal Cord Stimulation. A Verification of the Best Treatment Protocol
Brief Title: Burst Spinal Cord Stimulation for Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Sven Vanneste, Principal investigator, University Hospital, Antwerp
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: burst spinal cord stimulation
Record Dates: First submitted 2011-09-21; First posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Neuropathic Pain
Keywords: tonic, burst and placebo stimulation
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tonic (Experimental): 5 hz stimulation at an amplitude that the patient find bearable (+/- 1.5 mA)
  Interventions: Procedure: dorsal column stimulator
- Sham (Experimental): no stimulation, patient receive a sham stimulation (actually the IPG is not running)
  Interventions: Procedure: dorsal column stimulator
- burst (Experimental): 500 hz burst at 5 hz stimulation
  Interventions: Procedure: dorsal column stimulator

INTERVENTIONS:
Procedure: dorsal column stimulator — test different settings of stimulation
  Other Names: IPG is used by ST Jude medical together with an 88 lamitrode lead

SUMMARY:
Recently a novel stimulation design was developed, called burst stimulation. In a non-placebo controlled pilot study burst stimulation seemed superior to tonic stimulation over a period extending more than 2 years, and even though an incidental finding, this design seemed capable of suppressing pain without mandatory induction of paresthesias. This permits for the first time to scientifically prove that spinal cord stimulation is better than placebo stimulation. A study was therefore initiated to find out whether spinal cord stimulation is indeed capable of suppressing neuropathic limb pain in a placebo controlled way.

DETAILED DESCRIPTION:
Patients receive three type of stimulation (burst, tonic and sham). We want to compare these different stimulation protocol to verify which one is the one the patient prefer the most and have the least side-effects (paresthesia)

ELIGIBILITY:
All patients were selected after multidisciplinary discussion with a specialized pain physician, a psychological and psychiatric evaluation was performed to rule out psychogenic pain as well as other psychiatric morbidity contraindicating an implant. After authorization by the psychologist and psychiatrist an implant was offered.

Inclusion Criteria

* Patients enrolled in this study must meet the following inclusion criteria:
* Patients able to provide informed consent to participate in the study;
* Patient is between the age of 18 and 75;
* Patient has Failed Back Surgery Syndrome;
* Patient has a simulator implanted at the dorsal column spinal cord powered by an EON/EON Mini® internal pulse generator.
* Patient medication has remained stable for at least 4 weeks prior to baseline data collection;
* Patient agrees not to add or increase medication throughout the randomization trial period of the study;
* Patient is willing to cooperate with the study requirements including compliance with the treatment regimen and completion of all office visits.

Exclusion Criteria

A patient will be excluded from participation in this study if they meet any one of the following criteria:

* Patient has current evidence of any psychiatric disorder, as documented by the DSM-IV-TR criteria with psychotic characteristics;
* Patient has a history of life-threatening severe illness or is suffering from severe chronic disease other than the indication for the study;
* Patient has history of substance abuse or substance dependency in the past 6 months prior to baseline data collection;
* Patient currently participating in another clinical study;
* Patient with demand-type cardiac pacemakers, an infusion pump or any other implantable neurostimulator device except for the spinal cord stimulator under study;
* Patient is not willing to maintain current medication regimen;
* Female candidates of child bearing potential who are pregnant (confirmed by positive urine/blood pregnancy test), not using adequate contraception as determined by the investigator, or nursing (lactating) a child.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scales for pain back, pain limb, pain general and paresthesia

SECONDARY OUTCOMES:
VAS scores for pain now, worst pain, least pain and pain vigilance and awareness questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sven Vanneste, PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- University Hospital Antwerp, Edegem, Belgium

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473